CLINICAL TRIAL: NCT02442284
Title: An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With or Without Ribavirin (RBV) in US Veterans With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection (TOPAZ-VA)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With or Without Ribavirin in US Veterans With Genotype 1 Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-251
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis C; Cirrhosis; Hepatitis C Virus
Keywords: Chronic Hepatitis C; Interferon-Free; Hepatitis C Genotype 1; Hepatitis C Virus; Hepatitis C; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis; Hepatitis C | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3-DAA ± RBV for 12 or 24 weeks (Experimental): 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily] and dasabuvir [250 mg twice daily]) with or without weight-based ribavirin (± RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 or 24 weeks, dosed as per label based on genotype and presence of cirrhosis.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: Ribavirin — Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ombitasvir/paritaprevir/ritonavir and dasabuvir with or without ribavirin in US veterans with genotype 1 chronic hepatitis C virus infection.

ELIGIBILITY:
Inclusion Criteria:

* US military veteran currently receiving healthcare through the Veterans Health Administration
* Screening laboratory result indicating hepatitis C virus (HCV), genotype 1-infection
* Positive for hepatitis C antibodies or HCV RNA at least 6 months before Screening, and HCV RNA > 1,000 IU/mL at the time of Screening or HCV RNA > 1,000 IU/mL at the time of Screening with a liver biopsy consistent with chronic HCV-infection (or a liver biopsy performed prior to enrollment with evidence of chronic hepatitis C disease)

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Positive test result for hepatitis B surface antigen (HbsAg) or anti-HIV antibodies (HIV Ab)
* Prior or current use of any investigational or commercially available anti-HCV agents other than IFN, pegIFN, RBV or sofosbuvir
* Any current or past clinical evidence of Child-Pugh B or C classification
* Confirmed presence of hepatocellular carcinoma indicated on imaging techniques within 3 months prior to Screening or on an ultrasound performed at Screening for participants with cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2016-08-22 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Started | 99
Completed | 92
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Withdrew Consent | 2
Not completed — Lost to Follow-up | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (5.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. Participants with missing data after backwards imputation were imputed as nonresponders.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 99
percentage of participants | 93.9 [87.4 to 97.2]

2. Secondary Outcome: Percentage of Participants With Virologic Failure During Treatment
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment, or HCV RNA ≥ LLOQ at end of treatment.
Time Frame: up to 12 weeks (for 12-week treatment group) or up to 24 weeks (for 24-week treatment group
Population: Intent-to-treat (ITT) population: all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 99
percentage of participants | 1.0 [0.2 to 5.5]

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: All participants who received at least 1 dose of study drug, completed treatment, and had HCV RNA <LLOQ at the final treatment visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 99
percentage of participants | 2.2 [0.6 to 7.7]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12) Among Participants With Ongoing Psychiatric Disorders
Description: as for outcome 1
Time Frame: 12 weeks after the last actual dose of study drug
Population: All participants who received at least 1 dose of study drug (ITT population) and with ongoing psychiatric disorders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 48
percentage of participants | 95.8 [86.0 to 98.8]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks for participants treated for 12 weeks and up to 28 weeks for participants treated for 24 weeks).
Description: TEAEs and TESAEs are defined as any adverse event that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | 3-DAA ± RBV for 12 or 24 Weeks
Serious Adverse Events (participants affected / at risk) | 7/99
Other Adverse Events (participants affected / at risk) | 58/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA ± RBV for 12 or 24 Weeks (N=99)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
DRUG INTERACTION (General disorders) | 1
CHOLANGITIS (Hepatobiliary disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
SCHIZOPHRENIA (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA ± RBV for 12 or 24 Weeks (N=99)
ANAEMIA (Blood and lymphatic system disorders) | 5
DIARRHOEA (Gastrointestinal disorders) | 9
NAUSEA (Gastrointestinal disorders) | 15
FATIGUE (General disorders) | 28
OEDEMA PERIPHERAL (General disorders) | 5
HAEMOGLOBIN DECREASED (Investigations) | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
DIZZINESS (Nervous system disorders) | 8
HEADACHE (Nervous system disorders) | 20
ANXIETY (Psychiatric disorders) | 5
INSOMNIA (Psychiatric disorders) | 10
IRRITABILITY (Psychiatric disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.